

### **Clinical Study Protocol**

NCT Number: NCT05882279

Title: Evaluation of the Effectiveness of Risk Minimization Measures: A survey among pharmacists to assess the impact of the RMP material for patients on promoting the proper use of NINLARO in Japan

Study Number: C16065

Document Version and Date: Version 1.0 / 20-Apr-2023

Certain information within this document has been redacted (ie, specific content is masked irreversibly from view) to protect either personally identifiable information or company confidential information.



Version1.0: 20 April 2023



NON-INTERVENTIONAL SAFETY STUDY PROTOCOLOHICABLE TERRIPS OF LISE

uation of the Total State of the State of t Study title: Evaluation of the Effectiveness of Risk Minimization Measures: A survey among pharmacists to assess the impact of the RMP material for patients on promoting the proper use of NINLARO in Japan ?

Study number: C16065

Version number: Version 1.0 (20 April 2023)

Ethics statement: This study will be conducted in compliance with the protocol, the Declaration of Helsinki, International Society for Pharmacoepidemiology Guidelines for Good Epidemiology Practices, European Network of Centres for Pharmacoepidemiology and Pharmacovigilance Guidelines for Methodological Standards in Pharmacoepidemiology, Good Pharmacovigilance Practices, and all ale reproperty of Takeda applicable regulatory requirements.



Takeda C16065 NINLARO, ixazomib citrate

## Signature page

| NINLARO, ixazor | mib citrate | | , | |
|---|---|---|---|---|
| | Sig | nature page | | 150 |
| among pharma | | ness of Risk Minimization<br>act of the RMP material for<br>in Japan | Measures: A survey patients on | insofuse |
| Study numbe | r: C16065 | | < € | |
| | ber: Version 1.0 (20 April | , | dicaple | |
| Role | Head of Safety<br>Management, Global<br>Patient Safety | Printed Name | Director, Global Patient Safety Evaluation Japan, Takeda Development Center Japan Takeda Pharmaceutical Company Limited 1-1, Doshomachi 4- chome Chuo-ku, Osaka 540-8645, Japan | |
| Signature | non-comme | Date (DD-MMM-YYYY) | • | |

EU and UK QPPV:

| Vincilaan 7, 1930 |
|-------------------|
|-------------------|



Takeda C16065

Version1.0 : 20 April 2023

| C16065<br>NINLARO, ixazo | mih citrate | V | ersion1.0 : 20 April 2023 |
|---|---|---|---|
| NINEARO, IXAZO | This citrate | | Zaventem, Belgium Zaventem, Belgium Applicable Appl |
| Signature | | Date (DD-MMM-YYYY) | (SINSO) |
| | | | applice |
| | | * *C | "The |
| | | Ellifect | |
| | | is and | |
| | | ise offil | |
| | eicial, | | |
| | COMME | | |
| | of hours | | |
| 30. | | | |
| of Jakes | | | |
| operty | | | |
| Q.CO. | | | |



Version1.0 : 20 April 2023

# **Study information**

| Title | Evaluation of the Effectiveness of Risk Minimization Measures:<br>A survey among pharmacists to assess the impact of the RMP<br>material for patients on promoting the proper use of NINLARO<br>in Japan |
|---|---|
| Protocol number | C16065 |
| Protocol version identifier | 1.0 |
| Date of last version of protocol | Not Applicable |
| EU PAS register number | TBD |
| Active substance | ixazomib citrate (ATC code: L01XG03) |
| Medicinal product | NINLARO 2.3 mg hard capsules |
| | NINLARO 3 mg hard capsules |
| | NINLARO 4 mg hard capsules |
| Product reference | Not Applicable |
| Procedure number | Not Applicable |
| Joint PASS | No |
| Research question and objectives | The overall research question is to investigate whether the RMP material for patients (dosing instruction), which is defined as an additional risk minimization measure in J-RMP, is utilized for the proper use of NINLARO. |
| | Primary Objective: |
| 7.com | To assess the frequency of pharmacists who have provided patients with the contents of the RMP material for patients |
| ,00 | Secondary Objective: |
| Kot, | To assess the frequency of pharmacists who have obtained the RMP material for patients |
| regisi. For | To evaluate the depth of understanding of proper usage of NINLARO among pharmacists |
| Country(-ies) of study | Japan |
| Author | Global Patient Safety Evaluation Japan, Takeda Development<br>Center Japan |
| Marketing authorization holder(s) | TAKEDA PHARMACEUTICAL COMPANY LIMITED 1-1, Doshomachi 4-chome Chuo-ku, Osaka 540-8645, JAPAN |



Version1.0 : 20 April 2023

| MINEARO, MAZORIB CITALE | |
|---|---|
| MAH Contact Person | |
| MAIT CONTACT CISCH | |
| | Director, Global Patient Safety Evaluation Japan, Takeda |
| | Development Center Japan |
| | Takeda Pharmaceutical Company Limited |
| | Name of the second seco |
| | <sup>2</sup> 0, |
| | ::CO |
| | 0,1 |
| | ×O ~ |
| | :01 |
| | (0) |
| | 60, |
| | 29.3 |
| | M o |
| | S |
| | Me |
| c <sub>O</sub> | |
| 17,0 | |
| .,00 | |
| ₹0. | |
| 9.0 | |
| 100 | |
| <b>1</b> | |
| , O, | |
| (C) | |
| | Director, Global Patient Safety Evaluation Japan, Takeda Development Center Japan Takeda Pharmaceutical Company Limited |
| | Page 5 |



Takeda C16065

# Version1.0 : 20 April 2023

| TABI | LE O | F C | ON | TEN | ITS |
|------|------|-----|----|-----|-----|

| TAB | SLE OF ( | CONTENTS | 6 |
|---|---|---|---|
| 1.0 | | LIST OF ABBREVIATIONS | 8 |
| 2.0 | | RESPONSIBLE PARTIES | 9 |
| 3.0 | | ABSTRACT | 10 |
| 4.0 | | AMENDMENTS AND UPDATES | . 13 |
| 5.0 | | MILESTONES | 14 |
| 6.0 | | RATIONALE AND BACKGROUND RESEARCH QUESTION AND OBJECTIVES RESEARCH METHODS | 15 |
| 7.0 | | RESEARCH QUESTION AND OBJECTIVES | 15 |
| 8.0 | | RESEARCH METHODS | 16 |
| | 8.1 | STUDY DESIGN | 16 |
| | 8.2 | | |
| | | 8.2.1 Study population 8.2.2 Inclusion criteria 8.2.3 Exclusion criteria 8.2.4 Recruitment Process VARIABLES | 16 |
| | | 8.2.2 Inclusion criteria | 16 |
| | | 8.2.3 Exclusion criteria | 16 |
| | | 8.2.4 Recruitment Process | 16 |
| | 8.3 | VARIABLES | 17 |
| | 8.4 | DATA SOURCES | 17 |
| | 8.5 | DATA SOURCES | 18 |
| | 8.6 | DATA MANAGEMENT | 18 |
| | 8.7 | DATA ANALYSIS | 18 |
| | 8.8 | QUALITY CONTROL | 18 |
| | 8.9 | LIMITATIONS OF THE RESEARCH METHODS | 18 |
| 9.0 | | PROTECTION OF HUMAN SUBJECTS | 19 |
| | 9.1 | ETHICAL AND REGULATORY CONSIDERATIONS | 19 |
| | 9.2 | HCP INFORMATION AND CONFIDENTIALITY | 19 |
| 10.0 | ) | MANAGEMENT AND REPORTING OF ADVERSE EVENTS | 19 |
| | 10.1 | ADVERSE EVENTS | 19 |
| | 10.2 | SERIOUS ADVERSE EVENTS | 19 |
| 10 | 10.3 | Adverse Drug Reactions | 20 |
| | 10.4 | PRODUCT QUALITY COMPLAINTS | 20 |
| , | 10.5 | SPECIAL SITUATION REPORTS. | 20 |
| | 10.6<br>Produc | COLLECTION AND NOTIFYING OF ADVERSE EVENTS, SPECIAL SITUATION REPORTS AND CT QUALITY COMPLAINTS TO TAKEDA PHARMACOVIGILANCE | 21 |
| 11.0 | ) | PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS | 21 |



Properly of Takeda: For non-commercial use only and subject to the applicable Terms of use Takeda C16065 Version1.0: 20 April 2023



Takeda C16065 Version1.0 : 20 April 2023

NINLARO, ixazomib citrate

### **1.0 LIST OF ABBREVIATIONS**

| | Definition |
|---|---|
| | adverse drug reaction |
| | adverse event |
| | Company Core Data Sheet |
| CP | healthcare professional |
| D | ixazomib, lenalidomide and dexamethasone |
| | proteasome inhibitor |
| )C | product quality complaint |
| ИP | risk management plan |
| ИM | relapsed/refractory multiple myeloma |
| Æ | serious adverse event |
| )P | standard operating procedure |
| SR | special situation report |
| (akedai. Foi non.co | standard operating procedure special situation report The standard operating procedure special situation report The standard operating procedure special situation report |
| | QC<br>ИР<br>ИМ |



Takeda C16065 Version1.0 : 20 April 2023 NINLARO, ixazomib citrate

Subcontractor on survey implementation, Medilead, Inc. Tokyo Opera City Tower, 24F 3-20-2 Nishishinis-20-2 No. Septender of Lakeda. For non-comme



Takeda C16065 NINLARO, ixazomib citrate

#### 3.0 ABSTRACT

#### Title

reins of Use Evaluation of the Effectiveness of Risk Minimization Measures: A survey among pharmacists to assess the impact of the RMP material for patients on promoting the proper use of NINLARO in Japan

#### Rationale and background

Ixazomib (NINLARO) is an oral, highly selective, and reversible proteasome inhibitor (PI). Ixazomib preferentially binds and inhibits the chymotrypsin-like activity of the beta 5 subunit of the 20S proteasome. Ixazomib is administered as a citrate ester, designated ixazomib citrate. Ixazomib citrate, a prodrug, rapidly hydrolyses under physiological conditions to its biologically active form, ixazomib.

Ixazomib is approved in combination with lenalidomide and dexamethasone for the treatment of patients with relapsed/refractory multiple myeloma (rrMM) in a total of 72 countries worldwide as of 19 Nov 2022. In Japan, ixazomib is approved in combination with lenalidomide and dexamethasone for the indications of rrMM was approved on 30 Mar 2017 and was launched under the name of NINLARO on 24 May 2017. Each drug is dosed with different dosing schedules as follows:

- Ixazomib is dosed on Days 1, 8, 15 of a 28-day treatment cycle.
- Lenalidomide is dosed on Days 1 through 21 of a 28-day treatment cycle.
- Dexamethasone is dosed on Days 1, 8, 15, and 22 of a 28-day treatment cycle.

Overdose of ixazomib in combination with lenalidomide and dexamethasone (IRD therapy) has been reported in sponsored clinical trials, Investigator-Initiated Sponsored Research studies, and postmarking phase. Some of the overdoses have been associated with serious adverse events including multiple organ failure and death. Based on the safety signal evaluation of accidental overdose, overdose was endorsed as an identified risk of ixazomib. To minimize the risk of overdose, it is essential to ensure providers and patients understand the importance of adhering to the prescribed dosing schedule. The risk of overdose is described in Company Core Data Sheet (CCDS). As part of RMP in Japan (J-RMP), Takeda created the RMP material for patients to instruct the dosing of IRD therapy and has been distributed to patients via healthcare professional (HCP)s since its launch in Japan, in May 2017.

This web survey is planned to assess the effectiveness of distributed RMP material in prevention of ixazomib overdose in Japanese clinical practice.

#### Research question and objectives

The overall research question is to investigate whether the RMP material for patients (dosing instruction), which is defined as an additional risk minimization measure in J-RMP, is utilized for the proper use of NINLARO.

#### Primary Objective:

To assess the frequency of pharmacists who have provided patients with the contents of the RMP material for patients

#### Secondary Objective:

- To assess the frequency of pharmacists who have obtained the RMP material for patients
- To evaluate the depth of understanding of proper usage of NINLARO among pharmacists



Version1.0: 20 April 2023

## Study design

This web-based survey is intended for pharmacists who have instructed the dosing of IRD therapy to patients with rrMM. The survey will be self-administered via the web (i.e., the Internet). The questionnaires will be provided in Japanese.

#### **Population**

ermsofuse As most IRD therapy are prescribed as in-hospital prescriptions in Japan, in-hospital pharmacists are mainly involved in the explanation of how to take NINLARO in IRD therapy.

Pharmacists included in Nikkei Research Access Panel, active in clinical practice, and with valid contact details who meet the inclusion criteria, as listed in Section 8.2.2, will be randomly selected to participate in the survey.

#### Inclusion criteria

The survey will be conducted among pharmacists meeting the following inclusion criteria:

- Pharmacists who belong to hospitals prescribing NINLARO
- Pharmacists who have instructed the dosing of NINLARO in IRD therapy to patients

#### Exclusion criteria

None

#### **Variables**

In order to address the study objectives, the following information will be collected:

- Information on participating pharmacists (work experience, specialty)
- Information on hospitals where pharmacists are working (hospital type, number of beds/pharmacists, specialty)
- Information on the status of providing patients with the contents of the RMP material for patients
- Information on recollection of having obtained the RMP material for patients
- Information on pharmacists' awareness of the proper use of NINLARO
- Information on preferences for materials, etc.

#### **Data sources**

The survey is a primary data collection among pharmacists who have instructed the NINLARO dosing for IRD therapy to patients.

#### Study size

The sample size of 300 pharmacists was set. When n = 300, the width of the two-sided 95% confidence interval of the response ratio in the binary response questionnaire will be ± 5.7% at the maximum.



Takeda C16065 Version1.0: 20 April 2023

Adder the purple of Use only and subject to the applicable terms of Use only and subject to the applicable terms of Use only and subject to the applicable of Use only and Subject to the applicable o



| 1 20 April 2023 N/A N/A Initial protocol Reprints A pril 2023 N/A N/A Initial protocol Reprints A pril 2023 N/A N/A Initial protocol Reprints A pril 2023 N/A N/A Initial protocol | Takeda C16065 NINLARO, ixazomib clirate 4.0 AMENDMENTS AND UPDATES Number Date Section of study protocol Quadre Reason | Number | Date | Section of study protocol | Amendment or update | Reason |
|---|---|---|---|---|---|---|
| eubject to the applicable Term's | acommercial use only and subject to the applicable Terms | 1 | 20 April 2023 | N/A | N/A | Initial protocol |
| | T.commercial Use only and s | | | | cupiection | e applicable Len |



Version1.0 : 20 April 2023

### 5.0 MILESTONES

| Milestone | Planned date | Actual date | Comments | \s <sup>©</sup> |
|---|---|---|---|---|
| Start of data collection | June 2023 | <date></date> | <text></text> | |
| End of data collection | June 2023 | <date></date> | <text></text> | O <sup>1</sup> |
| Registration in the EU PAS register | May 2023 | <date></date> | <date></date> | ins |
| Study results | July 2023 | <date></date> | <text></text> | |

Property of Takeda: For non-commercial use only and subject to the admired the property of Takeda: For non-commercial use



 Takeda
 C16065
 Version1.0 : 20 April 2023

NINLARO, ixazomib citrate

#### **6.0 RATIONALE AND BACKGROUND**

Ixazomib is an oral, highly selective, and reversible PI. Ixazomib preferentially binds and inhibits the chymotrypsin-like activity of the beta 5 subunit of the 20S proteasome. Ixazomib is administered as a citrate ester, designated ixazomib citrate. Ixazomib citrate, a prodrug, rapidly hydrolyses under physiological conditions to its biologically active form, ixazomib.

Ixazomib is approved in combination with lenalidomide and dexamethasone for the treatment of patients with rrMM in a total of 72 countries worldwide as of 19 Nov 2022. In Japan, ixazomib is approved in combination with lenalidomide and dexamethasone for the indications of rrMM was approved on 30 Mar 2017 and was launched under the name of NINLARO on 24 May 2017. Each drug is dosed with different dosing schedules as follows.

- Ixazomib is dosed on Days 1, 8, 15 of a 28-day treatment cycle.
- Lenalidomide is dosed on Days 1 through 21 of a 28-day treatment cycle.
- Dexamethasone is dosed on Days 1, 8, 15, and 22 of a 28-day treatment cycle

Overdose of ixazomib in combination with lenalidomide and dexamethasone(IRD therapy) has been reported in sponsored clinical trials, Investigator-Initiated Sponsored Research studies, and post-market. Some of the overdoses have been associated with serious adverse events including multiple organ failure and death. Based on the safety signal evaluation of accidental overdose, overdose was endorsed as an identified risk of ixazomib. To minimize the risk of overdose, it is essential to ensure providers and patients understand the importance of adhering to the prescribed dosing schedule. The risk of overdose is described in CCDS. Takeda created the RMP material for patients to instruct the dosing of IRD therapy and has been distributed to patients via HCPs since the launch in Japan, in May 2017.

This web survey is planned to assess the effectiveness of distributed RMP material in prevention of ixazomib overdose in Japanese clinical practice.

# 7.0 RESEARCH QUESTION AND OBJECTIVES

The overall research question is to investigate whether the RMP material for patients (dosing instruction), which is defined as an additional risk minimization measure in J-RMP, is utilized for the proper use of NINLARO.

#### **Primary Objective:**

To assess the frequency of pharmacists who have provided patients with the contents of the RMP material for patients

#### Secondary Objective:

- To assess the frequency of pharmacists who have received the RMP material for patients
- To evaluate the depth of understanding of the proper use of NINLARO among pharmacists



Takeda C16065 NINLARO, ixazomib citrate

8.0 RESEARCH METHODS

#### 8.1 STUDY DESIGN

icable Terms of Use This web-based survey is intended for pharmacists who have instructed the dosing of IRD therapy to patients with rrMM. The survey will be self-administered via the web (i.e., the Internet). The questionnaires will be provided in Japanese.

#### 8.2 SETTING

#### 8.2.1 Study population

As most IRD therapy are prescribed as in-hospital prescriptions in Japan, in-hospital pharmacists are mainly involved in the explanation of how to take NINLARO in IRD therapy.

Pharmacists included in Nikkei Research Access Panel, active in clinical practice, and with valid contact details who meet the inclusion criteria, as listed in Section 8.2.2, will be randomly selected to participate in the survey.

8.2.2 Inclusion criteria

The survey will be conducted among pharmacists meeting the following inclusion criteria:

- Pharmacists who belong to hospitals prescribing NINLARO
- Pharmacists who have instructed the dosing of NINLARO in IRD therapy to patients
  - 8.2.3 Exclusion criteria

None

#### 8.2.4 Recruitment Process

Recruitment will be conducted as follows:

- Based on the information from the Nikkei Research Access Panel, pharmacists working in hospitals with experience in prescribing NINLARO will be invited to participate in the survey via email and portal site, in accordance with local requirements. The survey background and objectives, the contact information for questions, the intended use of data, and the proposed compensation will be explained to the pharmacists at this step.
- If the pharmacists agree to participate in the survey, they will access the link for the web questionnaire and answer it following the instructions. If the questionnaire is started but not yet completed, the pharmacist will be sent a reminder by e-mail.



Takeda C16065 NINLARO, ixazomib citrate

#### 8.3 VARIABLES

, applicable Terms of Use In order to address the study objectives, the following information will be collected (all questionnaires using options):

- Information on participating pharmacists
  - Work experience
  - Specialty (with or without licenses related to cancer therapy)
- Information on hospitals where pharmacists are working
  - Hospital type
  - Number of beds
  - Number of pharmacists
  - Specialty (with or without cancer central hospitals designation)
- Information on the status of providing patients with the contents of the RMP material for patients
  - Status of providing patients with NINLARO dosing schedule
  - For pharmacists who provide patients with NINLARO dosing schedule, materials that have been used for explanation
- Information on recollection of having obtained the RMP material for patients
- Information on pharmacists' awareness of the proper use of NINLARO
  - Understanding of the proper NINLARO dosing schedule
  - Understanding of the importance of providing NINLARO dosing schedule
- Information on preferences for materials, etc.
  - Self-perceived awareness of RMP for NINLARO
  - Factors to look for in materials for patient
  - Preferred media (paper / electronic)

#### 8.4 DATA SOURCES

The survey is a primary data collection among pharmacists who have instructed the NINLARO dosing for IRD therapy to patients. Sampling will be done based on the information from Nikkei Research Access Panel. Potential respondents will be invited to participate in the survey via e-mail and portal site, in accordance with local requirements. If the pharmacists agree to participate in the survey, they will access the link for the web questionnaire in the e-mail or "my page" on the portal site and answer the questionnaire following the instructions. The data will be collected in a web questionnaire, which will be filled in by the participating pharmacist.



Takeda C16065 NINLARO, ixazomib citrate

8.5 STUDY SIZE

reins of Use The sample size (the targeted final analysis set) of 300 pharmacists was set. When n = 300, the width of the two-sided 95% confidence interval of the response rate in the binary response questionnaire will be ± 5.7% at the maximum.

#### 8.6 DATA MANAGEMENT

Data collection will be carried out by Medilead, Inc. via web questionnaire in accordance with their applicable standard operating procedures (SOPs). Collected data will be entered and stored in a secure server for this survey. The statistical analysis will be conducted using ASSUM. to the ac

#### 8.7 DATA ANALYSIS

The baseline characteristics of participants will be summarized.

For each question, the number and/or percentage of participants who responded for each answer option is calculated. Cross-tabulations are also performed between participants' backgrounds and/or questions, as appropriate.

#### 8.8 QUALITY CONTROL

Medilead, Inc, will create the raw data set (data cleaning), cross-tabulation tables, and survey result report, according to their procedures.

#### 8.9 LIMITATIONS OF THE RESEARCH METHODS

The potential for selection bias of pharmacists participating in a survey is an inherent bias/limitation to any study based on volunteer participation. In this study, sampling will be done based on the information from the Nikkei Research Access Panel. It doesn't include all pharmacists working in hospitals with experience in prescribing NINLARO so that the generalization and external validity of the results is restricted. In addition, participants have to be willing (and able) to answer a questionnaire online. These pharmacists may not be fully representative of the whole targeted population (1).

In terms of exposure bias, pharmacists may have potential conflicts of interest with the survey.

Recall bias is minimized through broad sampling to include respondents with varying lengths of exposure to the RMP material and having experience in prescribing NINLARO.

Pharmacists will be allowed to participate only once. The format will allow for the questionnaire to be started but saved and completed at another time. Thus, stakeholder bias or unverified respondents are not applicable. A Reminder will be sent by e-mail to both non-responders and those who started but not yet completed to reduce non-response bias.

Web surveys may promote social desirability bias which refers to the tendency of pharmacists to give socially desirable/expected responses instead of choosing those reflecting their current knowledge or behavior. Social desirability can affect the validity of survey research findings regarding the knowledge



Takeda C16065 Version1.0: 20 April 2023

NINLARO, ixazomib citrate

of both RMP and the proper usage of NINLARO, but the use of prepopulated items in the questionnaire ins of Use could reduce this bias (2).

#### 9.0 PROTECTION OF HUMAN SUBJECTS

The survey is non-interventional. HCP information such as name and e-mail address will not be linked in any way to the answers provided by the HCPs and all answers will be anonymous to the study sponsor. Data collected will remain absolutely confidential, and only aggregated data will be analyzed and communicated in a report.

#### 9.1 ETHICAL AND REGULATORY CONSIDERATIONS

The survey will follow the regulatory and ethical requirements in Japan.

The objective of this study is not to influence physicians' prescribing behaviour by any means.

#### 9.2 HCP Information and Confidentiality

Persons participating in the study will be informed of the targets of the investigation, the intended use of data, and recipients of these data. The answers provided will be collected in an anonymous way.

Data will be recorded in a central database and will include security elements to prevent others than authorized staff from accessing data.

#### MANAGEMENT AND REPORTING OF ADVERSE EVENTS 10.0

#### 10.1 **ADVERSE EVENTS**

An adverse event (AE) is any untoward medical occurrence in a patient administered a medicinal product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (for example, an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to this medicinal product.

#### SERIOUS ADVERSE EVENTS

A serious adverse event (SAE) is any untoward medical occurrence that at any dose:

- Results in death
- Is life-threatening (NOTE: The term "life-threatening" in the definition of "serious" refers to an event/reaction in which the patient was at risk of death at the time of the event/reaction; it does not refer to an event/ reaction which hypothetically might have caused death if it were more severe)
- Requires inpatient hospitalization or results in prolongation of existing hospitalization
- Results in persistent or significant disability/incapacity



Takeda C16065 Version1.0 : 20 April 2023

NINLARO, ixazomib citrate

- Is a congenital anomaly/birth defect
- Is a medically important event

Medical and scientific judgment should be exercised in deciding whether other situations should be considered serious such as important medical events that might not be immediately life-threatening or result in death or hospitalisation but might jeopardise the patient or might require intervention to prevent one of the other outcomes listed in the definition above. Examples of such events are intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalization, or development of drug dependency or drug abuse.

#### 10.3 ADVERSE DRUG REACTIONS

An Adverse Drug Reaction (ADR) is "a response to a medicinal product which is noxious and unintended." Response in this context means that a causal relationship between a medicinal product and an adverse event is at least a possibility.

#### 10.4 PRODUCT QUALITY COMPLAINTS

A Product Quality Complaint (PQC) is any written, electronic, or oral communication that alleges deficiencies related to the identity, quality, durability, reliability, safety, strength, purity, effectiveness, or performance of a product or device and combination product after it is released for distribution.

# 10.5 SPECIAL SITUATION REPORTS

A Special Situation Report (SSR) includes any of the following events:

- Pregnancy: Any case in which a pregnancy patient is exposed to a Takeda Product or in which
  a female patient or female pattner of a male patient becomes pregnant following treatment with
  Takeda Product. Exposure is considered either through maternal exposure or via semen
  following paternal exposure
- Breastfeeding: Infant exposure from breast milk
- Overdose: All information of any accidental or intentional overdose
- Drug abuse, misuse, or medication errors: All information on medicinal product abuse, misuse or medication error (potential or actual)
- Gathering detailed information for AEs occurring in the pediatric or elderly population, as described in GVP Module VI
- Lack of efficacy of Takeda product
- Accidental/Occupational exposure
- Use outside the terms of the marketing authorization, also known as "off-label"

Information on the below situations, if received, should be collected and transmitted to GPSE (PV) although they are not considered special situations per GVP Module VI:

Suspected transmission of an infectious agent: All information on a suspected (in the sense of



Takeda C16065 Version1.0: 20 April 2023

NINLARO, ixazomib citrate

confirmed or potential) transmission of an infectious agent by a medicinal product.

- Use of falsified / counterfeit medicinal product
- Drug-drug interactions and drug-food interactions
- Inadvertent or accidental exposure with or without an AE

A SSR should be reported even if there is no associated AE.

# reins of Use COLLECTION AND NOTIFYING OF ADVERSE EVENTS, SPECIAL SITUATION 10.6 REPORTS AND PRODUCT QUALITY COMPLAINTS TO TAKEDA PHARMACOVIGILANCE

Safety events spontaneously notified to the investigator(s) or research team

If during the conduct of the study the investigator(s) or a member of the research team is spontaneously informed by a HCP or patient of an SAE, AE, ADR, SSR or PQC where the event/complaint pertains to a Takeda product (or unbranded generic), such information should be notified to the relevant Takeda Pharmacovigilance department within 1 working day for fatal or lifethreatening SAEs, within 4 calendar days for other SAEs, and within 7 calendar days for all other events. As such reports are spontaneously notified, causality of any adverse events should be assumed unless there is evidence to the contrary.

- AE reports and SSRs shall be reported to
- PQCs shall be reported to

# 11.0 PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS

Study results will be submitted possibly for publication in a peer-review journal.

#### 12.0 REFERENCES

- (1) Wyatt JC. When to use web-based surveys. J Am Med Inform Assoc 2000; 7(4):426-9.
- Alethod. 10. Method. 10. Metho (2) Nederhof AJ. Methods of coping with social desirability bias: A review. Eur. J. Soc. Psychol. 1985;



| | Document | | | |
|---|---|---|---|---|
| Number<br>1 | Version 1.0 | Date 20 April | Title NINLARO RMM Effectiveness | 01 |
| | | 2023 | Study_Questionnaire | ) |
| | | | Yo. | |
| | | | 204 | |
| | | | *No | |
| | | | 40 | |
| | | | C. C | |
| | | | . 17. | |
| | | | a suloie | |
| | | | and subject | |
| | | | 4 and subject | |
| | | orl | y and subject | |
| | | Seoli | A and subject | |
| | . ( | aluse on | y and subject | |
| | Ċ | AUSEON | y and subject | |
| | melici's | aluseon | y and sulpies | |
| | ominerci | aluseon | y and sulpies | |
| | . r.commerci | aluseon | y and subject | |
| | , on cominerci | alle of | y and sulpies | |
| | or non-commerci | AUSEON | y and sulpies | |
| | For non-commerci | aluseon | y and sulpies | |
| 200 | kot vourcounture, con vource, | allse of | y and subject | |
| Heda | For non-commerci | Allseor | y and subject | |
| Kakeda | kot non commerci | AUSON | yand sulpies | |
| ofTakeda | kot hourouthinetci, | Aluseon | y and subjection of the subjec | |
| of the da | For hon-commerci | Allseor | y and subjection of the subjec | |
| sperty of Takeda | For non-commerci | Aluseor | Title NINLARO_RMM Effectiveness Study_Questionnaire Admittable Territe Nandesthie Attacher Admittable Territe Nandesthie | |